CLINICAL TRIAL: NCT06547944
Title: A Phase 1b Clinical Study of Lenalidomide in Combination With Zanubrutinib and Obinutuzumab (ZGR) in the Treatment of Newly Diagnosed Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) With Therapeutic Indications
Brief Title: Zanubrutinib, Obinutuzumab and Lenalidomide in Newly Diagnosed Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Acronym: ZGR in TN CLL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023063
Record Dates: First submitted 2024-07-28; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Newly Diagnosed
Keywords: Zanubrutinib; Lenalidomide; Obinutuzumab; newly diagnosed CLL/SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib; Lenalidomide; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZGR regimen (Experimental): Dose Escalation lenalidomide combined with Zanubrutinib and Obinutuzumab (Dose escalation will occur using a 3+3 design)
  Recommended phase II dose (RP2D) lenalidomide combined with Zanubrutinib and Obinutuzumab
  Interventions: Drug: Zanubrutinib; Drug: Lenalidomide; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Zanubrutinib — 160mg bid/d, from C1 to CR and MRD-negative or C24
Drug: Lenalidomide — From C3 dose escalation, all 3 dose groups climbed from 5 mg/d to 10 mg/d, 15 mg/d, and 20 mg/d respectively, Taking 21 days of medication and 7 days of rest, 1 cycle every 28 days to CR and MRD-negative or C24
Drug: Obinutuzumab — 1000 mg C1, d1/d8/15; 1000 mg C2-6, d1

SUMMARY:
The ZGR regimen limited-course regimen was designed to combine three targeted agents, zanubrutinib, obinutuzumab (a third-generation CD20 monoclonal antibody), and lenalidomide, to deepen the depth of remission in patients with new-diagnosis CLL/SLL, with a view to achieving the goal of discontinuation of the drug and long-term remission after discontinuation of the drug, and prolonging the PFS, and at the same time, the regimen no longer includes cytotoxic chemotherapeutic agents, such as fludarabine and cyclophosphamide, which improves the CLL/ SLL patients' treatment tolerance, and can eliminate the treatment limitation for elderly or poorly tolerated CLL/SLL patients.

DETAILED DESCRIPTION:
BTK inhibitor monotherapy for CLL/SLL can obtain 80-90% ORR and give patients long-term survival, but most patients only obtain PR efficacy, even after up to 7-8 years of continuous treatment, the proportion of patients with CR can only be improved from less than 10% to about 30%, and it is very difficult for any patient to achieve MRD negativity, so it is determined that the mode of treatment of BTK inhibitor monotherapy is long-term continuous administration for tumor control. In order to change this pattern of long-term continuous treatment, and to shorten the long-term continuous treatment to a limited cycle of treatment, it is necessary to deepen the depth of remission by combining the treatment with other mechanisms of drugs, or even to achieve MRD-negativity in order to realize the discontinuation of the drug.

Lenalidomide is an oral immunomodulatory drug with direct antitumor effects and indirect antitumor effects by acting on a variety of immune cells in the tumor microenvironment. Lenalidomide alone, in combination with CD20 monoclonal antibody (rituximab), or (and) BTK inhibitors for the treatment of R/R CLL/SLL has shown therapeutic responses, with the best response to triple therapy of lenalidomide in combination with rituximab and BTK inhibitors. combination therapy showed the best response.

The ZGR limited-course regimen that combines zanubrutinib, obinutuzumab, and lenalidomide in the treatment of patients with primary diagnosis of CLL/SLL, which can deepen the depth of remission, with a view to achieving the goal of discontinuation of the drug and long-term remission after discontinuation of the drug, and prolonging the PFS, and at the same time, the regimen are removed cytotoxic chemotherapeutic agents, such as fludarabine, to increase the tolerance of the treatment in patients with CLL/SLL, and can eliminate the need for treatment of elderly or poorly tolerated patients with CLL/SLL. treatment limitations in poorly tolerated CLL/SLL patients.

ELIGIBILITY:
Inclusion Criteria:

* 1） Patients were not categorized by gender ，Age ≥18;
* 2） Confirmed diagnosis of CLL or SLL;
* 3）Patients must be untreated, or not undergoing standardized treatment for the first time, under the following conditions:
* a) Not treated with fludarabine-containing or bendamustine-containing or rituximab-containing regimens;
* b) Have not been treated with the application of chlorambucil, or have applied chlorambucil for less than 4 weeks (alone or in combination with adrenal glucocorticoids);
* (c) If the above treatment has been applied, it must be stopped for 2 weeks before enrollment in the group to start the treatment.
* 4） Indications for treatment of CLL/SLL include, inter alia (at least one of the following conditions is met)

  1. Evidence of progressive bone marrow failure: as evidenced by progressive decrease in hemoglobin and/or platelets;
  2. Giant spleen (e.g., >6 cm below the left costal margin) or symptomatic splenomegaly;
  3. Giant lymph node enlargement (e.g., longest diameter >10 cm) or symptomatic lymph node enlargement;
  4. Progressive lymphocytosis, e.g., >50% lymphocytosis within 2 months, or lymphocyte doubling time (LDT) <6 months. When initial lymphocytes are <30 x 10^9/L, LDT alone cannot be used as a therapeutic indication;
  5. CLL/SLL resulting in symptomatic organ dysfunction (e.g., skin, kidney, lung, spine, etc.)
  6. Autoimmune hemolytic anemia (AIHA) and/or immune thrombocytopenia (ITP) that does not respond well to corticosteroids or other standard therapy;
  7. Presence of at least one of the following disease-related symptoms: i) weight loss ≥10% without apparent cause within the previous 6 months; ii) severe fatigue (e.g., ECOG physical status ≥2; inability to perform routine activities); iii) temperature >38°C for ≥2 weeks without evidence of infection; iv) nocturnal night sweats for >1 month without evidence of infection;
* 5） ECOG≤2
* 6) Major organ function within 7 days prior to treatment, meet the following criteria: routine blood test criteria: platelets ≥30×10^9/L; biochemical tests need to meet the following criteria: total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤2.5 ULN; creatinine clearance ≥ 30 ml/min; and cardiac Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ low limit of normal (50%);
* 7) Male and female patients of childbearing age agree to use reliable contraception throughout the study period and for 4 weeks after the end of study treatment;
* 8) Patients need to have an expected survival of ≥ 6 months;
* 9) Patients need to voluntarily participate in this study by signing an informed consent form.

Exclusion Criteria:

* Patients who met any of the following criteria were excluded from the study:
* (1) Malignancies other than CLL/SLL (including active CNS lymphoma) have been diagnosed or treated within the past year;
* (2) There has been clinical evidence of Richter transformation;
* (3) Non-lymphoma-related hepatic and renal impairment: alanine aminotransferase (ALT) > 3 times the upper limit of normal, alanine transaminase (AST) > 3 times the upper limit of normal, total bilirubin (TBIL) > 2 times the upper limit of normal, and serum creatinine clearance < 30 ml/min;
* (4) Other serious medical disorders that would interfere with the study (e.g., uncontrolled diabetes mellitus, gastric ulcers, grade 3 or 4 atrial fibrillation or persistent atrial fibrillation of any grade, other serious cardiorespiratory diseases, etc.). The judgmental decision is vested in the investigator;
* (5) Patient who had infected with Human Immunodeficiency Virus (HIV) or active Hepatitis B Virus (HBV) infection, or any uncontrolled active systemic infection requiring intravenous antibiotics;
* (6) Clinically manifested CNS dysfunction or invasion of the center;
* (7) Patients who have undergone a major surgical procedure (excluding lymph node biopsy) within the last 14 days or who require a major surgical procedure in anticipation of treatment;
* (8) Inability to swallow capsules or suffering from malabsorption syndromes, disorders significantly affecting gastrointestinal function, having undergone gastric or small bowel resection, symptomatic inflammatory bowel disease or ulcerative colitis, and partial or complete intestinal obstruction.
* (9) Requires treatment with potent cytochrome P450 (CYP) 3A inhibitors;
* (10) Pregnant or lactating women of childbearing age who are not using contraception;
* (11) Patients with clinically significant cardiovascular abnormalities (New York Heart Association (NYHA) classification: III/IV), myocardial infarction within 6 months prior to enrollment, malignant arrhythmias (including QTC ≥ 480 ms), poorly controlled blood pressure (systolic ≥ 150 mmHg, diastolic ≥ 100 mmHg) despite the use of antihypertensive medications, and uncontrolled angina;
* (12) Persistent uncontrolled bleeding;
* (13) History of life-threatening hemorrhage, especially from irreversible causes;
* (14) Need for high doses of several anticoagulants that cannot be briefly discontinued;
* (15) Thrombotic events within three months of treatment initiation;
* (16) Patients with severe hypersensitivity to the active ingredient of the study drug or to any of its excipients;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of lenalidomide in combination regimens were determined in newly diagnosed CLL/SLL patients, | From the date of first dose of study drugs until RP2D was determined(Approximately 4 months)]
The incidence, nature and severity of adverse events (AE) were determined according to NCI-CTCAE v5.0 evaluation criteria | From first dose to 30 days after the last dose of Zanubrutinib or lenalidomide or Obinutuzumab

SECONDARY OUTCOMES:
overall response rate(ORR) | From first dose to 30 days after the last dose of Zanubrutinib or lenalidomide or Obinutuzumab
  Defined as the proportion of patients assessed as CR, CRi, or PR according to the IWCLL 2018 criteria at or before initiation of subsequent antitumor therapy.
overall survival Overall survival(OS) | Up to 5 years
  Defined as the time interval from enrollment to death for patients in an intentional-treatment population (ITT). If the patient continues to survive or if his or her life is unknown, the date of death will be the nearest point in time when the patient is known to be alive.
Progress-free survival(PFS) | Up to 5 years
  Defined as the time interval from enrollment to disease progression or death of a patient in an intention-to-treat population (ITT), whichever comes first. For those who did not progress at the time of exit or whose time to disease progression was not recorded, the last examination date was used as the end date.
Duration of tumor remission(DOR) | Up to 5 years
  Defined as the time interval between first recorded disease remission and first recorded evidence of PD in patients in an intention-to-treat population (ITT). No progression or time to disease progression was recorded at the time of exit from the trial, with the date of last examination as the end date.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tam CS, Brown JR, Kahl BS, Ghia P, Giannopoulos K, Jurczak W, Simkovic M, Shadman M, Osterborg A, Laurenti L, Walker P, Opat S, Chan H, Ciepluch H, Greil R, Tani M, Trneny M, Brander DM, Flinn IW, Grosicki S, Verner E, Tedeschi A, Li J, Tian T, Zhou L, Marimpietri C, Paik JC, Cohen A, Huang J, Robak T, Hillmen P. Zanubrutinib versus bendamustine and rituximab in untreated chronic lymphocytic leukaemia and small lymphocytic lymphoma (SEQUOIA): a randomised, controlled, phase 3 trial. Lancet Oncol. 2022 Aug;23(8):1031-1043. doi: 10.1016/S1470-2045(22)00293-5. Epub 2022 Jul 7. PMID 35810754
- [Background] Ferrajoli A, Lee BN, Schlette EJ, O'Brien SM, Gao H, Wen S, Wierda WG, Estrov Z, Faderl S, Cohen EN, Li C, Reuben JM, Keating MJ. Lenalidomide induces complete and partial remissions in patients with relapsed and refractory chronic lymphocytic leukemia. Blood. 2008 Jun 1;111(11):5291-7. doi: 10.1182/blood-2007-12-130120. Epub 2008 Mar 11. PMID 18334676
- [Background] Badoux XC, Keating MJ, Wen S, Lee BN, Sivina M, Reuben J, Wierda WG, O'Brien SM, Faderl S, Kornblau SM, Burger JA, Ferrajoli A. Lenalidomide as initial therapy of elderly patients with chronic lymphocytic leukemia. Blood. 2011 Sep 29;118(13):3489-98. doi: 10.1182/blood-2011-03-339077. Epub 2011 Jul 1. PMID 21725050
- [Background] Badoux XC, Keating MJ, Wen S, Wierda WG, O'Brien SM, Faderl S, Sargent R, Burger JA, Ferrajoli A. Phase II study of lenalidomide and rituximab as salvage therapy for patients with relapsed or refractory chronic lymphocytic leukemia. J Clin Oncol. 2013 Feb 10;31(5):584-91. doi: 10.1200/JCO.2012.42.8623. Epub 2012 Dec 26. PMID 23270003
- [Background] Ujjani C, Wang H, Skarbnik A, Trivedi N, Ramzi P, Khan N, Cheson BD. A phase 1 study of lenalidomide and ibrutinib in combination with rituximab in relapsed and refractory CLL. Blood Adv. 2018 Apr 10;2(7):762-768. doi: 10.1182/bloodadvances.2017015263. PMID 29610115